CLINICAL TRIAL: NCT02041403
Title: MAY RENAL RESISTIVE INDEX BE AN EARLY PREDICTIVE TOOL OF POST-OPERATIVE COMPLICATIONS IN MAJOR SURGERY?
Brief Title: RENAL RESISTIVE INDEX POST-OPERATIVE COMPLICATIONS IN MAJOR SURGERY?
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: CE ICH-158/12
Record Dates: First submitted 2014-01-18; First posted 2014-01-22 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Major High Risk Operations; Renal Resistive Index; Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal resistive Index

SUMMARY:
An observational trial aiming to verify whether does any relationship exist between renal resistive index and postoperative outcome in major high risk surgery

DETAILED DESCRIPTION:
Renal resistive index was measured just after major high risk operations and then patients were observed searching for any surgical and medical-related complications during the first post-operative week

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* major surgical operations

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to major high risk surgery
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Complications | 7 post-operative days
  Recording any postoperative complication occurred within the first postoperative week

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Giustiniano, MD, Principal Investigator — Humanitas Research Hospital -Dept. Anesthesia and Intensive Care
Locations (2):
- Italy (2):
  - Sant'Ambrogio Clinical Institute - Cardiac Anesthesia Unit, Milan, Milano
  - Humanitas Research Hospital - Dept. Anesthesia and Intensive Care Unit, Rozzano, Milano